CLINICAL TRIAL: NCT06271538
Title: A Randomized Double-Blind Placebo-controlled Clinical Trial on the Efficacy of Skål Pro (Lactobacillus Plantarum 299 and Galacto-oligosaccharides) in Improving Severity of Symptoms, Stool Forms, Quality of Life and Psychological Dysfunction in Patients With Irritable Bowel Syndrome (IBS)
Brief Title: Evaluation of Efficacy of Skål Pro Powder on Symptoms of Irritable Bowel Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: EP Plus Group Sdn Bhd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP-USM-122023-001
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Syndrome; Gastrointestinal Diseases; Colonic Diseases, Functional; Intestinal Disease; Digestive System Disease; Pathologic Processes; Colonic Disease; Disease
Keywords: probiotic; Lactobacillus plantarum 299v; randomized controlled study
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases; Colonic Diseases, Functional; Intestinal Diseases; Digestive System Diseases; Pathologic Processes; Colonic Diseases; Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Skal Pro (Experimental): Skal Pro in the form of 2g sachet powder contains 10 billion CFU of freeze-dried Lactobacillus plantarum 299v (LP299V) and galactooligosaccharides (GOS).
  Interventions: Combination Product: Skal Pro
- Placebo (Placebo Comparator): Placebo is an oral formulation of inert powder. Placebo and Skal Pro are identical in shape, size, colour, packaging and taste.
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Skal Pro — One sachet Skal Pro per day containing Lactobacillus plantarum 299v 1x10^10 CFU and GOS
  Arms: Skal Pro
Other: Placebo — One sachet per day identical in shape, size, colour, packaging and taste to the Skal Pro sachet
  Arms: Placebo

SUMMARY:
The objective of this randomized, double-blind, placebo-controlled study is to evaluate the effectiveness of Skal Pro in alleviating symptoms, enhancing stool consistency, improving quality of life, and addressing psychological distress in individuals diagnosed with irritable bowel syndrome (IBS), as compared to those who receive no intervention.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a condition linked to disturbances in the gut-brain axis and dysbiosis. Although probiotic modulation of dysbiosis appears promising for IBS treatment, identifying the specific beneficial strains remains uncertain. Furthermore, even with an effective probiotic strain, variations in efficacy among populations are observed due to environmental heterogeneity, particularly dietary influences.

This study seeks to provide efficacy insights into Skal Pro powder 2g (containing Lactobacillus plantarum 299v 1x10^10 colony forming unit (CFU) and GOS), shedding light on the unique mechanisms of LP299V within the Malaysian population through a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* IBS diagnosed using the Rome IV criteria
* Age above 18 years old and any gender
* Any subtypes of IBS (diarrhea, constipation or mixed)

Exclusion Criteria:

* Presence of red flag symptoms (weight loss, anemia, night symptoms, abdominal mass, strong family history of cancer)
* Was prescribed antibiotic (s) within the past one month
* Medical conditions that contraindicate probiotic use including severe sepsis and pregnancy
* Presence of bowel malignancy
* Diagnosis of bowel infection within the past one month
* Previous abdominal surgeries
* Patients with overt psychiatric illnesses including schizophrenia and manic disorders
* A history of allergy to probiotic
* Was prescribed probiotic (s) within the past one month
* Was previously prescribed probiotic Skal Pro™ (LP299V™)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Improving the severity of symptoms in individuals with IBS, assessed by IBS Symptom Severity Scale (IBSSSS) | Assessed at baseline, Week 1, Week 2, and Week 4.
  IBSSS questionnaire contains five questions that measures, on a 100-point visual analogue scale (VAS), the severity of abdominal pain, the frequency of abdominal pain, the severity of abdominal distension, dissatisfaction with bowel habits, and interference with quality of life (QOL). All five components contribute to the scores equally, yielding a theoretically range of 0 - 500, with a higher score indicating worse condition. The Malay version questionnaire will be used.

SECONDARY OUTCOMES:
Change in stool consistency (Bristol Stool Scale), assessed by daily stool diary | Assessed daily from baseline to Week 4.
  Daily diary of stool consistency of each bowel movement based on Bristol Stool Scale (Type 1-7), from type 1-2 = separate hard lump stool, type 3-4= ideal stool, type 5-7 =loose stool
Change in stool frequency and satisfaction after passing stool, assessed by daily stool diary | Assessed daily from baseline to Week 4.
  Daily diary of number of bowel movements.
Change in abdominal bloating, assessed by Bloating Severity Questionnaire (BSQ) | Assessed at baseline, Week 1, Week 2, and Week 4.
  Originally developed by Thiwan et al., this research group then translated and validated the BSQ in the Malay language (BSQ-M) [13]. There are 2 sub-scales, the 6-item Sev-Gen (Severity-General) and 5-item Sev-24 (Severity-24 hour) with responses in seven-point Likert scale on different degree of severity (from 1 = never to 7=always). For this study, only the Sev-Gen will be used.
Improvement in Quality of Life, assessed by EQ-5D-5L Questionnaire | Assessed at baseline, Week 1, Week 2, and Week 4.
  The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009, and consist of 2 sections, 1) the EQ-5D descriptive system and 2) the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain or discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health the participant can imagine' and 'The worst health the participant can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. The Malay version questionnaire will be used.
Change in Visceral Sensitivity Index | Assessed at baseline, Week 1, Week 2, and Week 4.
  The Visceral Sensitivity Index (VSI) is a 15-item questionnaire which measures gastrointestinal symptom-specific anxiety. Replies to each item are provided on a 6-point scale from "strongly disagree" (scored as 0) to "strongly agree" (scored as 5). A Malay version of the questionnaire was developed using standard forward-back translation procedures. The Malay version questionnaire will be used.
Assessment of psychological dysfunction suing Catastrophizing Questionnaire | Assessed at baseline, Week 1, Week 2, and Week 4.
  The Coping Strategies Questionnaire (CSQ) - Catastrophizing (CAT) subscale consists of six questions on a 6-point Likert scale, with response options ranging from 0 (never) to 5 (very frequently). The Malay version questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Yeong Yeh Lee, MD, PhD, Principal Investigator — Hospital Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No